CLINICAL TRIAL: NCT04097522
Title: Neurofeeback for Chronic Pain Project (NFB Project)
Brief Title: The Effectiveness of Neurofeedback for the Treatment of Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Collaborators: TIYGA Health (Unknown)
Responsible Party: Principal Investigator, Anthony Jones, Clinical Professor, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 244779
Record Dates: First submitted 2018-11-21; First posted 2019-09-20 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain
Keywords: neurofeedback
MeSH Terms: conditions — Chronic Pain | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: Half of the participants that take part in the neurofeedback procedures will receive sham neurofeedback, whilst the other half will receive neurofeedback from an area the investigators believe to be associated with increasing pain resilience. Participants may or may not receive sham neurofeedback, and will be made aware of this fact.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A number of the studies include double-blind neurofeedback, where half of the participants receive sham neurofeedback, and half receive actual neurofeedback from a region thought to increase pain resilience. The experimenter, participant, and care provider will all be blinded as to which condition the participant is in until the participant leaves the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real neurofeedback (Active Comparator): Participants receive neurofeedback from a region of the brain thought to be associated with increasing pain resilience
  Interventions: Other: Neurofeedback
- sham neurofeedback (Sham Comparator): Participants receive neurofeedback from a region of the brain thought to be unrelated with increasing pain resilience
  Interventions: Other: Neurofeedback

INTERVENTIONS:
Other: Neurofeedback — During the neurofeedback intervention, participants will be shown visual representations of their own brain activity in real-time. Over a number of sessions participants will teach themselves to increase this brain activity, in order to increase their own pain resilience levels.

SUMMARY:
This study evaluates the effectiveness of neurofeedback (teaching participants to gain control over their own brainwaves) in chronic pain. The study is made up of four pilot studies. Participants who take part will undergo the cold pressor test, submerging their hand in cold water in order to simulate chronic pain. Brain activity will be measured using electroencephalography (EEG).

DETAILED DESCRIPTION:
Chronic pain is a persisting pain which often exists in the absence of detectable tissue damage. It is also associated with feelings of depression, anxiety, and despair. Current treatments for chronic pain usually involves drug treatments, which often has unwanted side effects.

This study aims to assess the effectiveness of neurofeedback, which refers to teaching participants to gain control over their own brainwaves, as an intervention to treat chronic pain. It is believed that by teaching participants to gain control over a brain signal associated with pain resilience, the participant can reduce some of the negative effects associated with chronic pain.

Participants who take part in this study will have their brain activity recorded using electroencephalography (EEG), and have pain elicited using the cold pressor test (CPT), which involves the participant submerging their wrist in cold water to elicit a chronic pain-like sensation. This is a safe, regularly used method, and the participant is free to remove their hand early if the pain becomes too great.

Some participants who take part will undergo neurofeedback training, which will involve them viewing a signal associated with pain resilience, and learning to increase it over multiple sessions.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Must be aged 40 or older

Exclusion Criteria:

* Current or planned hospitalisation during the period of study.
* Non-English speaking participants
* Participants already involved in clinical trials, if it is not possible to schedule around this
* Unable, in the opinion of the research investigator, to comply or adhere to the requirements of the study.
* Patients with chronic pain in both upper limbs
* History of brain injury, stroke or neurosurgical procedures
* An implanted neurostimulator (e.g., deep brain stimulator)
* Damaged skin tissue on the head, or a skin condition such as severe eczema, or any skin allergies
* Failure of cognitive test (Montreal Cognitive Assessment) will exclude participants from taking part in studies that use neurofeedback procedures
* Some but not all of the study will be unavailable to participants currently undergoing psychotherapy (such as cognitive behavioural therapy).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-10-05 (Estimated); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Changes in pain ratings | Throughout the participant's time in the study, approximately 8-16 weeks. (16 sessions which occur approximately twice per week,depending on participant's availability.).
  The investigators will monitor changes in pain ratings, which are ratings of current pain level, given on a scale from 0-10 using a Visual Analogue Scale (VAS). These ratings will be given by participants while undergoing the experimental procedures in the study.

SECONDARY OUTCOMES:
Smartphone app measures of changes in of chronic pain-related symptoms | Throughout the participant's time in the study, an average of 12 weeks.
  Participants may be given a smartphone app with which to record their current chronic pain levels using sliders. The sliders have no units, sliding towards maximum will indicate high chronic pain, sliding towards minimum indicates low chronic pain. Participants will be free to choose whether to use this or not.
Changes in brain activity caused by neurofeedback procedures | Throughout the participant's time in the study, an average of 12 weeks.
  The investigators will monitor changes in brain activity associated with neurofeedback procedures, measured using EEG (focusing on the alpha band). It is expected that neurofeedback will cause an increase in brain activity associated with pain resilience.
Self-report: participant's own ratings of pain experienced | through study completion, an average of 12 weeks.
  Participant will self-report on their own levels of pain experienced, using a visual analogue scale (VAS) from 0 (no pain) to 10 (worst pain imaginable).
Questionnaire: Brief Pain Inventory | through study completion, an average of 12 weeks.
  Participant self-assesses current or recent pain using a scale which ranges from from 0 (no pain/does not interfere) to 10 (worst pain imaginable/completely interferes), with high scores representing a worse outcome.
Questionnaire: Participant Demographics | Administered at initial session, one day only
  General information about participant's age, gender, etc
Questionnaire: EQ5D (developed by EuroQol group) | through study completion, an average of 12 weeks.
  General measure of overall health, includes a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state), with 0 representing the worst outcome
Questionnaire: Hospital Anxiety and Depression Scale | through study completion, an average of 12 weeks.
  Participant self-reports feelings of anxiety and depression, ticking against responses representing their current feelings.
Questionnaire: McGill Short Form | through study completion, an average of 12 weeks.
  Questionnaire assessing participants current pain level
Questionnaire: Medical history | Administered at initial session, one day only
  Participant notes current medications and previous major operations
Assessment: Montreal Cognitive Assessment | through study completion, an average of 12 weeks.
  Used to assess participant's cognitive abilities, several questions are answered verbally or by writing on the form
Questionnaire: Pain Catastrophizing Scale | through study completion, an average of 12 weeks.
  Measures the extent to which a person 'catastrophises' i.e. overly worries about a pain or events associated with pain, and includes a scale ranging from 0 (Not at all) to 4 (all the time), with high scores for negatively phrased events representing the worst outcomes
Questionnaire: PANAS (Positive and Negative Affect Schedule) | through study completion, an average of 12 weeks.
  Participant rates a number of words which describe different feelings and emotions, and includes a scale ranging from 1 (Very slightly or not at all) to 5 (Extremely), with high scores for negatively phrased events representing the worst outcomes
Questionnaire: PSEQ (Pain Self-Efficacy Questionnaire) | through study completion, an average of 12 weeks.
  Participant rates how confident they are that they can do the following things at present, despite their current pain. Scale ranges from 0 (not confident at all) to 6 (completely confident), with a high score indicating confidence in one's own ability to cope or perform a task despite the pain
Assessment: Tender Points Survey | through study completion, an average of 12 weeks.
  Assessor gently but firmly presses a finger against certain pressure points on the participant to asses levels of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Salford Royal NHS Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
No individually identifiable participant data will be shared outside of the research group, and the University of Manchester (for the purposes of audit).
  Non-identifiable (pseudo-anonymised) data will be shared with TIYGA Health through their phone app if participants choose to upload this information, however, no phone location data, names, ore any other personal information will be shared with them. Participants are free to choose not to use the phone app with no penalties for not taking part
Time Frame: Non-identifiable information will be shared, only when participants choose to share it during the neurofeedback training sessions (8-16 weeks). TIYGA Health will retain the data in line with GDPR (General Data Protection Regulation) requirements for pseudo-anonymised data - retaining data for 5 years before deletion (after last data entry), and may archive accounts if no new data is added for 2 years
Access Criteria: Please contact us at james.henshaw-2@manchester.ac.uk and we will provide email access to the full DMP (Data Management Plan, available at link below)
URL: https://dmponline.dcc.ac.uk/plans/29612